CLINICAL TRIAL: NCT04558567
Title: A Phase 4, Open-Label, Single-Arm Study to Evaluate the Effects of Vogelxo(R) on 24-hour Ambulatory Blood Pressure Monitoring in Hypogonadal Men Using Therapeutic Testosterone Replacement Therapy
Brief Title: Vogelxo(R) ABPM Study in Hypogandal Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Upsher-Smith Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P361-502
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism | interventions — Testosterone Propionate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label (Other)
  Interventions: Drug: Vogelxo

INTERVENTIONS:
Drug: Vogelxo — 50mg (1 tube, 5g gel) to 100mg (2 tubes, 10g gel)

SUMMARY:
A Phase 4 ABPM study in Hypogonadal Men

DETAILED DESCRIPTION:
A single-arm, open-label, uncontrolled study consisting of a 4-week screening phase, 4-week titration phase, and 16-week treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male whose age is between 18 and 80 years, inclusive, at the time of screening.
2. Considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead electrocardiogram (ECG) results, and physical examination findings at screening.
3. Meets the study definition of clinical hypogonadism, as evidenced by serum testosterone concentrations:

   1. Two serum testosterone concentrations < 300 ng/dL collected in the morning (between 0630 hours and 1000 hours local time) on at least 2 days separated by a minimum of 48 hours.
   2. Presence of at least 1 sign or symptom that may be related to low testosterone values and is/are consistent with hypogonadism
4. Naïve to testosterone replacement, clomiphene, compounded or over-the-counter androgenic steroid derivatives and dehydroepiandrosterone, including investigational products that may affect the reproductive hormonal system within the past 2 months.
5. Willingness and the ability to apply topical testosterone gel as instructed by the study staff and comply with the requirements of this study protocol.
6. Intact skin surfaces on the upper arms and shoulders where the topical testosterone will be applied.

Exclusion Criteria:

1. Two testosterone concentrations < 100 ng/dL during screening.
2. Prolactin concentration > 1 x upper limit of normal (ULN).
3. Current or recurrent ulcer, erosion, lichenification, inflammation psoriasis, eczema or use of topical corticosteroids on the upper arms and shoulders. Tattoo application or removal in the region of study drug application.
4. Known skin intolerance to alcohol or allergy to any of the ingredients of the study drug.
5. History of treatment with growth hormone, anti-estrogen or estrogen treatment within 90 days prior to screening.
6. Currently taking glucocorticoids > 7.5 mg prednisone equivalent per day (eg, hydrocortisone 30 mg, methylprednisolone 6 mg, or dexamethasone 1.2 mg) for 1 week before SV1 and through Day 1, and any use of opioids within 5 half-lives prior to Day 1.
7. Currently taking, unstable doses within 14 days prior to first administration of study drug or anticipated to receive any antihypertensive medications, over-the-counter medications, supplements or herbal medicines known to affect blood pressure during study participation. These medications or supplements include diet pills (eg, phenylpropanolamine, sibutramine), nasal decongestants (eg, phenylephrine hydrochloride, pseudoephedrine, naphazoline hydrochloride), certain stimulants (eg, amphetamine, methylphenidate dexmethylphenidate, dextroamphetamine), monoamine oxidase inhibitors (MAO), atypical antipsychotics (eg, clozapine, olanzapine).
8. History of prostate (current or in the past) or breast cancer.
9. Severe lower urinary tract symptoms as indicated by an International Prostate Symptom Score (I-PSS) > 19.
10. Prostate-specific antigen (PSA) > 3.0 ng/mL; men treated with 5-alpha reductase inhibitors (eg, dutasteride, finasteride) are eligible for participation as long as PSA levels are not > 1.5 ng/mL.
11. Body mass index > 50 kg/m2.
12. Sitting SBP < 80 mm Hg and > 150 mm Hg or sitting DBP < 50 mm Hg and > 100 mm Hg at any point during screening.
13. HbA1c > 11% at screening.
14. A current condition, therapy, laboratory abnormality, history of clinically significant medical or psychiatric conditions or other circumstance or reasons which, in the opinion of the investigator or the study staff, might pose a risk to the subject, make participation not in the subject's best interest, confound the results of the study (eg, if subject cannot comply with requirements of the study), make the subject an unsuitable candidate to receive study drug, or interfere with the subject's participation for the full duration of the study.
15. History, suspicion, or evidence of significant drug or alcohol abuse or illicit steroid use within the previous 12 months prior to screening, as determined by the investigator.
16. The subject is a smoker or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 6 months before the first dose of study drug.
17. Clinical laboratory analysis shows any of the following abnormal results:

    * Hematocrit > 50%
    * Alanine aminotransferase or aspartate aminotransferase > 3 × ULN
18. Severe or end-stage chronic kidney disease documented by eGFR < 30 mL/min.
19. Subject works night shifts.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the 24-hour ABPM average SBP | 20 weeks
  Average SBP will be calculated from ABPM measurements taken twice each hour over the 24-hour period. An ABPM measurement session will be standardized and performed during on-site clinic visits at baseline (before treatment) and on the last day of treatment (week 20) to minimize subject variability.

SECONDARY OUTCOMES:
Change from baseline in 24-hour average diastolic blood pressure (DBP) | 20 weeks
Change from baseline in 24-hour average heart rate (HR) | 20 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Upsher-Smith Clinical Trial Site #6, Birmingham, Alabama
  - Upsher-Smith Clinical Trial Site #2, Anaheim, California
  - Upsher-Smith Clinical Trial Site #1, Miami, Florida
  - Upsher-Smith Clinical Trials Site #7, Garden City, New York
  - Upsher-Smith Clinical Trials Site #4, North Charleston, South Carolina
  - Upsher-Smith Clinical Trials Site #5, San Antonio, Texas
  - Upsher-Smith Clinical Trials Site #8, San Antonio, Texas